CLINICAL TRIAL: NCT02776124
Title: A Randomized Phase II Trial to Assess the Effect of Oral Supplements on the Nutritional Status of Locally Advanced Nasopharyngeal Carcinoma Patients During Concurrent Chemotherapy
Brief Title: Effect of Oral Supplements on the Nutritional Status of Locally Advanced Nasopharyngeal Carcinoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Collaborators: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Zhu, Professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1405135-4
Record Dates: First submitted 2016-05-03; First posted 2016-05-18 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nutritional status; nasopharyngeal carcinoma; Nutritional Counseling; concurrent chemoradiotherapy; oral nutritional supplements
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ONS group (Experimental): Individualized dietary counseling+ONS(Healing elements)during CRT Interventions: (Healing elements)
  Interventions: Dietary Supplement: Healing Elements,Methuselah Medical Technology
- control group (No Intervention): Individualized dietary counseling during CRT

INTERVENTIONS:
Dietary Supplement: Healing Elements,Methuselah Medical Technology — ONS group will receive Healing Elements ONS everyday during CRT
  Arms: ONS group

SUMMARY:
Malnutrition is very common in locally advanced nasopharyngeal carcinoma(NPC) patients undergoing current chemoradiotherapy (CRT) due to dysphagia, mucositis, nausea and other treatment-related problems. Malnutrition is associated with lower physical functioning, lower immune status, more severe (grade III/IV) late RT-induced toxicities, treatment interruption of chemo(radio)therapy, lower chemotherapy response rates, hospital readmission, impaired quality of life (QoL), and increased mortality. Although the international guidelines recommend early nutritional support in the presence of nutritional risk, the best type of nutritional intervention is still unclear. Individualized dietary counseling showed beneficial effects in nutritional intake, nutritional status and QoL in head and neck cancer patients undergoing RT or CRT-treatment; oral nutritional supplements (ONS) was most acceptable in Chinese NPC patients. Previous nutritional intervention trials in head-neck cancer patients have been conducted on small samples and did not clarify the role of oral nutritional supplements (ONS). Accordingly, although current guidelines recommend as grade A the use of ONS associated with dietary counseling for head-neck cancer patients undergoing RT, the efficacy of this nutritional intervention still needs to be evaluated in adequately sized and randomized clinical trials for Chinese NPC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed、pathologically proven nasopharyngeal carcinoma（Stage III/IV）
2. Concurrent radiation and chemotherapy(platinum )
3. Karnofsky score over 60
4. No evidence of metastatic disease
5. No significant cardiac, chest, gastrointestinal or renal morbidities

Exclusion Criteria:

1. age <18 years
2. ongoing artificial nutrition
3. refusal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-08 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Body weight(kg)change during concurrent chemotherapy | every week during the course of radiotherapy, up to 6-7 weeks

SECONDARY OUTCOMES:
Disease-free survival | 2 years
  From date of randomization until date of first documented disease progression or death from any cause, assessed up to 2 years.
Score of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Core 35 (EORTC QLQ-HN35) during the concurrent treatment | every 2 weeks during the course of radiotherapy, up to 6-7 weeks
  participants will be followed for the duration of hospital stay, an expected average of 6-7 weeks
Number of participants with treatment-related adverse events as assessed by CTCAE v3.0 | every week during the course of radiotherapy, up to 6-7 weeks
Body cell mass(kg) change measured by multifrequency segmental bioelectrical impedance analysis | every week during the course of radiotherapy, up to 6-7 weeks
Fat mass (kg) change measured by multifrequency segmental bioelectrical impedance analysis | every week during the course of radiotherapy, up to 6-7 weeks
Fat free mass (kg) change measured by multifrequency segmental bioelectrical impedance analysis | every week during the course of radiotherapy, up to 6-7 weeks
Skeletal muscle mass (kg) change measured by multifrequency segmental bioelectrical impedance analysis | every week during the course of radiotherapy, up to 6-7 weeks
Phase angle(°) change measured by multifrequency segmental bioelectrical impedance analysis | every week during the course of radiotherapy, up to 6-7 weeks
Serum albumin（g/L) change | every 2 weeks during the course of radiotherapy, up to 6-7 weeks
Serum prealbumin（mg/dL) change | every 2 weeks during the course of radiotherapy, up to 6-7 weeks
Serum transferrins（mg/dL）change | every 2 weeks during the course of radiotherapy, up to 6-7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided